CLINICAL TRIAL: NCT00700661
Title: A Multicenter, Double-Blind, Placebo-Controlled, Randomized, Parallel-Group, Study to Determine the Efficacy of Montelukast in the Treatment of Exacerbations in Asthmatic Patients Aged 2-to-5 Years
Brief Title: A Study of MK0476 in the Treatment of Asthma Patients Aged 2-5 Years (0476-907)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0476-907; MK0476-907; 2007_572
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Drug
  Interventions: Drug: montelukast
- 2 (Placebo Comparator): Pbo
  Interventions: Drug: placebo (unspecified)

INTERVENTIONS:
Drug: montelukast — One montelukast 4-mg chewable tablet (CT) administered once daily at bedtime. Duration of Treatment: 48 Weeks
  Other Names: MK0476; SINGULAIR ®
  Arms: 1
Drug: placebo (unspecified) — Matching-image Montelukast placebo. Duration of Treatment: 48 Weeks
  Arms: 2

SUMMARY:
A study to determine the efficacy of MK0476 in the Treatment of Asthmatic Patients Aged 2 to 5 Years.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female between and including the ages of 2 and 5 years
* Patient was treated with steroids for an asthma episode in the last 3 months
* Patient was admitted to the hospital or emergency room in the last 3 months
* Patient is able to chew a tablet

Exclusion Criteria:

* Patient has been in a research study in the past 4 weeks
* Patient has visited the emergency room for an asthma episode in the past week
* Patients has a history of stomach, heart, liver, nerve, kidney or blood disease

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Actual)
Dates: Start 2001-01; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
asthma episodes in 2 - 5 year old children | at 12 months

SECONDARY OUTCOMES:
the number of treatments and duration of asthma episodes | at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Bisgaard H, Zielen S, Garcia-Garcia ML, Johnston SL, Gilles L, Menten J, Tozzi CA, Polos P. Montelukast reduces asthma exacerbations in 2- to 5-year-old children with intermittent asthma. Am J Respir Crit Care Med. 2005 Feb 15;171(4):315-22. doi: 10.1164/rccm.200407-894OC. Epub 2004 Nov 12. PMID 15542792